CLINICAL TRIAL: NCT01192139
Title: Bioequivalence Study of the Fixed Dose Combination of 5 mg Saxagliptin and 500 mg Metformin XR Tablet (Manufactured in Mt Vernon, IN) Relative to 5 mg Saxagliptin Tablet and 500 mg Metformin XR Tablet (Manufactured in Evansville, IN) Coadministered to Healthy Subjects in a Fed Condition
Brief Title: Bioequivalence Study of the Fixed Dose Combination of 5 mg Saxagliptin and 500 mg Metformin XR Tablet (Manufactured in Mt Vernon, IN) Relative to 5 mg Saxagliptin Tablet and 500 mg Metformin XR Tablet (Manufactured in Evansville, IN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-111
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg saxagliptin + a single 500 mg metformin XR tablet (Experimental)
  Interventions: Drug: saxagliptin; Drug: metformin XR
- FDC tablet (5 mg saxagliptin + 500 mg metformin XR) (Fed) (Experimental): under fed state
  Interventions: Drug: saxagliptin + metformin XR (FDC tablet)
- FDC tablet (5 mg saxagliptin + 500 mg metformin XR) (Fasting) (Experimental): under fasted state
  Interventions: Drug: saxagliptin + metformin XR (FDC tablet)

INTERVENTIONS:
Drug: saxagliptin — Tablets, Oral, 5 mg, once daily, Single dose
  Other Names: Onglyza
  Arms: 5 mg saxagliptin + a single 500 mg metformin XR tablet
Drug: metformin XR — Tablets, Oral, 500 mg. once daily, Single dose
  Other Names: Glucophage XR
  Arms: 5 mg saxagliptin + a single 500 mg metformin XR tablet
Drug: saxagliptin + metformin XR (FDC tablet) — Tablet, Oral, (saxagliptin 5 mg)(metformin XR 500 mg), once daily, Single dose
  Arms: FDC tablet (5 mg saxagliptin + 500 mg metformin XR) (Fasting); FDC tablet (5 mg saxagliptin + 500 mg metformin XR) (Fed)

SUMMARY:
The purpose of this study is to demonstrate bioequivalence (BE) of a 5 mg saxagliptin/500 mg metformin extended release (XR) fixed-dose combination (FDC) tablet (manufactured in Mt Vernon, Indiana [IN]) to coadministered 5 mg saxagliptin and 500 mg metformin XR tablet (manufactured in Evansville, IN) in fed healthy subjects.

DETAILED DESCRIPTION:
This study is designed to evaluate if the FDC tablet of 5 mg saxagliptin/500 mg metformin extended release (manufactured in Mt Vernon, Indiana) is bioequivalent to the coadministered 5 mg saxagliptin and 500 mg metformin XR tablet (manufactured in Evansville, Indiana)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECG), and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive
* Ages 18 to 45, inclusive

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Major surgical procedure within 4 weeks prior to randomization
* Positive serology test for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Clinically significant history or presence of any of the following conditions: heart, liver, or kidney disease, neurologic or psychiatric disease
* History of gastrointestinal disease within the past 3 months
* Any clinically significant medical condition that could potentially affect your participation in the study and/or personal well-being, as judged by the investigator
* Donated blood or blood products to a blood bank, blood transfusion or participated in a clinical study (except a screening visit) requiring withdrawal of blood within 4 weeks prior to randomization
* Unable to tolerate oral and/or intravenous (IV) medications
* Unable to tolerate the puncturing of veins for drawing of blood
* Known allergy or hypersensitivity to any component of the study medication
* History of any significant drug allergies (such as anaphylaxis or hepatotoxicity)
* Used any prescription drugs or over the counter products to control acid (for example, Prevacid, Mylanta or Rolaids) within 4 weeks prior to randomization
* Used any other drugs including over the counter medications and herbal preparations within 1 week prior to randomization
* Taken any investigational drug or placebo (inactive drug) within 4 weeks prior to randomization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- [Derived] Boulton DW, Smith CH, Li L, Huang J, Tang A, LaCreta FP. Bioequivalence of saxagliptin/metformin extended-release (XR) fixed-dose combination tablets and single-component saxagliptin and metformin XR tablets in healthy adult subjects. Clin Drug Investig. 2011;31(9):619-30. doi: 10.2165/11590290-000000000-00000. PMID 21819160
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent screening evaluations to determine eligibility within 21 days before dosing, and were admitted to the clinical facility the evening before dosing (Day -1). On Day 1 of Period 1, a total of 30 participants who met all of the inclusion and none of the exclusion criteria were randomly assigned to 1 of 6 treatment sequences.
Groups:
- Treatment Sequence ABC: Treatment A (period 1): 5 mg saxagliptin + a single 500 mg metformin XR tablet; Treatment B (period 2): fixed-dose combination (FDC) Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions; Treatment C (period 3): FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions. Participants underwent at least a 3-day washout period between each treatment.
- Treatment Sequence ACB: Treatment A (period 1): 5 mg saxagliptin + a single 500 mg metformin XR tablet; Treatment C (period 2): FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions; Treatment B (period 3): fixed-dose combination (FDC) Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions. Participants underwent at least a 3-day washout period between each treatment.
- Treatment Sequence BAC: Treatment B (period 1): fixed-dose combination (FDC) Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions; Treatment A (period 2): 5 mg saxagliptin + a single 500 mg metformin XR tablet; Treatment C (period 3): FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions. Participants underwent at least a 3-day washout period between each treatment.
- Treatment Sequence BCA: Treatment B (period 1): fixed-dose combination (FDC) Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions; Treatment C (period 2): FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions; Treatment A (period 3): 5 mg saxagliptin + a single 500 mg metformin XR tablet. Participants underwent at least a 3-day washout period between each treatment.
- Treatment Sequence CAB: Treatment C (period 1): FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions; Treatment A (period 2): 5 mg saxagliptin + a single 500 mg metformin XR tablet; Treatment B (period 3): fixed-dose combination (FDC) Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions. Participants underwent at least a 3-day washout period between each treatment.
- Treatment Sequence CBA: Treatment C (period 1): FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions; Treatment B (period 2): fixed-dose combination (FDC) Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions; Treatment A (period 3): 5 mg saxagliptin + a single 500 mg metformin XR tablet. Participants underwent at least a 3-day washout period between each treatment.
Period: Period 1
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled and Treated Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White | 17
  Black or African American | 12
  Asian | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 21
Height [Mean (Standard Deviation); unit: cm] | 170.0 (9.22)
Weight [Mean (Standard Deviation); unit: kg] | 78.31 (13.74)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.97 (3.07)

OUTCOME MEASURES:

1. Primary Outcome: Saxagliptin Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf])
Description: Area under the plasma concentration versus time curve from time 0 extrapolated to infinity; calculated as AUC0-t [calculated using the linear trapezoidal rule] + Ct/Kel, where Ct was the last measurable concentration and Kel was the terminal rate constant
Time Frame: Periods 1, 2, and 3 (samples taken before dosing, and at 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 36 and 48 hours after dosing)
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Treatment A - Saxagliptin + Metformin XR, Fed: 5 mg saxagliptin tablet + a single 500 mg metformin XR tablet under fed conditions
- Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed: fixed-dose combination (FDC) tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions
- Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting: FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*hr/mL | 107.28 (25.13) | 111.72 (26.55) | 103.35 (23.15)
Statistical Analysis 1: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed vs Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; If there was no difference between the bioavailabilities of saxagliptin from the FDC tablet versus saxagliptin from coadministration of a saxagliptin tablet and a metformin XR tablet under fed conditions, then 24 subjects would have provided 99% power to conclude bioequivalence (BE) with respect to Cmax and AUC0-inf. If there was a 5% difference, then 24 subjects would have provided 94% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within 0.800 to 1.250 for both Cmax and AUC0-inf of saxagliptin; Ratio of Geometric Least Squares Means = 1.039, 90% CI 2-sided [1.011 to 1.068] — Ratio=Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed vs Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Test type: Non-Inferiority or Equivalence — Lack of food effect was concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within (80%, 125%) for both Cmax and AUC(INF) of saxagliptin and metformin; Ratio of Least Squares Means = 1.078, 90% CI 2-sided [1.049 to 1.108] — Ratio=Treatment B/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed; Geometric least squares means for treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 104.65
Statistical Analysis 4: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Geometric least squares means for treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 108.74
Statistical Analysis 5: Comparison: Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Geometric least squares mean for treatment C; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 100.84

2. Secondary Outcome: Saxagliptin Terminal Half-life (T1/2)
Description: terminal half life; calculated as ln(2)/Kel
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
hours | 8.46 (2.85) | 8.56 (3.04) | 9.21 (3.91)

3. Secondary Outcome: Saxagliptin Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-t])
Description: Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration (Ct), calculated using the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*hr/mL | 105.47 (24.98) | 109.88 (26.36) | 101.52 (23.01)
Statistical Analysis 1: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed vs Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Test type: Superiority or Other; Ratio of Geometric Least Squares Mean = 1.039, 90% CI 2-sided [1.011 to 1.068] — Ratio = Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed vs Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 1.080, 90% CI 2-sided [1.051 to 1.110] — Ratio=Treatment B/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed; Geometric least squares mean for treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 102.84
Statistical Analysis 4: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Geometric least squares mean for treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 106.89
Statistical Analysis 5: Comparison: Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Geometric least squares mean for treatment C; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 98.99

4. Primary Outcome: Saxagliptin Observed Maximum Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 26.84 (8.26) | 27.25 (7.95) | 28.85 (8.62)
Statistical Analysis 1: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed vs Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 1.021, 90% CI 2-sided [0.940 to 1.109] — Ratio=Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed vs Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Test type: Non-Inferiority or Equivalence — Lack of food effect was concluded if the fed to fasted ratios of geometric means were entirely contained within (80%, 125%) for both Cmax and AUC(INF) of saxagliptin; Ratio of Geometric Least Squares Means = 0.949, 90% CI 2-sided [0.873 to 1.031] — Ratio = Treatment B/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed; Geometric least squares mean for treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 25.68
Statistical Analysis 4: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Geometric least squares mean for treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 26.21
Statistical Analysis 5: Comparison: Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Geometric least squares mean for treatment C; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 27.63

5. Secondary Outcome: Time to Achieve the Observed Maximum Saxagliptin Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
hours | 1.65 (0.65) | 1.48 (0.75) | 0.65 (0.50)

6. Secondary Outcome: Saxagliptin Fraction of AUC(0-inf) Contributed by AUC(0-t) (AUC[0-t]/AUC[0-inf])
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ratio | 0.983 (0.006) | 0.983 (0.006) | 0.982 (0.008)

7. Secondary Outcome: Active Metabolite BMS-510849 AUC(0-inf)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*hr/mL | 291.72 (79.21) | 295.94 (75.40) | 289.06 (66.89)

8. Secondary Outcome: Active Metabolite BMS-510849 AUC(0-t)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*hr/mL | 284.46 (78.25) | 289.03 (74.80) | 281.79 (65.91)

9. Secondary Outcome: Active Metabolite BMS-510849 Cmax
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 49.71 (16.94) | 49.28 (14.59) | 49.09 (15.46)

10. Secondary Outcome: Active Metabolite BMS-510849 T1/2
Description: terminal half life; calculated as ln(2)/Kel
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
hours | 13.88 (1.53) | 13.65 (1.72) | 14.04 (1.33)

11. Secondary Outcome: Active Metabolite BMS-510849 Tmax
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
hours | 2.38 (0.76) | 2.42 (0.88) | 1.46 (0.70)

12. Secondary Outcome: Active Metabolite BMS-510849 AUC(0-t)/AUC(0-inf)
Time Frame: Period 1 (samples taken before dosing, and at 0.167,0.25,0.5,0.75,1,1.5,2,3,4,5,6,7,8,10,12,18,24,36 and 48 hours after dosing)
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ratio | 0.974 (0.008) | 0.975 (0.008) | 0.974 (0.006)

13. Primary Outcome: Metformin AUC(0-inf)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Treated participants (the smaller sample size for AUC[0-inf] was due to the inability to estimate potassium chloride for some participants)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 25 | 24 | 23
ng*hr/mL | 5865.92 (2357.15) | 5516.97 (2423.08) | 5073.70 (1406.45)
Statistical Analysis 1: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed vs Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; If there was no difference between the bioavailabilities of metformin from the FDC tablet versus metformin from coadministration of a saxagliptin tablet and a metformin XR tablet under fed conditions, then 24 subjects would have provided 99% power to conclude BE with respect to Cmax and AUC0-inf. If there was a 5% difference, then 24 subjects would have provided 96% and 97% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — BE concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within (80%, 125%) for both Cmax and AUC(INF) of saxagliptin and metformin; Ratio of Least Squares Geometric Means = 0.915, 90% CI 2-sided [0.836 to 1.002] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed vs Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Test type: Non-Inferiority or Equivalence — lack of food effect concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within (80%, 125%) for both Cmax and AUC(INF) of saxagliptin and metformin; Ratio of Geometric LS Mean and 90% CI = 1.010, 90% CI 2-sided [0.918 to 1.111] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed; Geometric least squares means for treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 5542.2
Statistical Analysis 4: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Geometric least squares mean for treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 5072.9
Statistical Analysis 5: Comparison: Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Geometric least squares mean for treatment C; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 5023.3

14. Secondary Outcome: Metformin AUC(0-t)
Description: as for outcome 3
Time Frame: as for outcome 12
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*hr/mL | 5617.39 (2181.99) | 5200.46 (2203.34) | 4896.95 (1340.41)
Statistical Analysis 1: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed vs Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Test type: Superiority or Other; Ratio of Geometric Least Squares Mean = 0.920, 90% CI 2-sided [0.854 to 0.992] — Ratio=Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed vs Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 1.025, 95% CI 2-sided [0.951 to 1.105] — Ratio=Treatment B/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed; Geometric least squares means for treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 5287.1
Statistical Analysis 4: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Geometric least squares mean for treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 4866.2
Statistical Analysis 5: Comparison: Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Geometric least squares means for treatment C; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 4746.8

15. Primary Outcome: Metformin Cmax
Time Frame: as for outcome 1
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 629.73 (160.14) | 586.87 (150.63) | 657.23 (187.67)
Statistical Analysis 1: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed vs Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; If there was no difference between the bioavailabilities of metformin from the FDC tablet versus metformin from coadministration of a metformin XR tablet under fed conditions, then 24 subjects would have provided 99% power to conclude BE with respect to Cmax and AUC0-inf. If there was a 5% difference, then 24 subjects would have provided 96% and 97% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within 0.800 to 1.250 for both Cmax and AUC0-inf of metformin; Ratio of Geometric Least Squares Means = 0.933, 95% CI 2-sided [0.865 to 1.007] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed vs Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of Geometric Least Squares Means = 0.898, 90% CI 2-sided [0.832 to 0.969] — Ration = Treatment B/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - Saxagliptin + Metformin XR, Fed; Geometric least squares mean for treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 608.41
Statistical Analysis 4: Comparison: Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed; Geometric least squares mean for treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 567.85
Statistical Analysis 5: Comparison: Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting; Geometric least squares mean for treatment C; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 632.39

16. Secondary Outcome: Metformin T1/2
Description: terminal half life; calculated as ln(2)/Kel
Time Frame: Period 1 (before dosing, 0.167,0.25,0.5,0.75,1,1.5,2,3,4,5,6,7,8,10,12,18,24,36 and 48 hours after dosing)
Population: Treated participants (the smaller sample size for T1/2 was due to the inability to estimate Kel for some of the subjects).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 25 | 24 | 23
hours | 10.7 (5.90) | 12.6 (7.05) | 14.9 (7.40)

17. Secondary Outcome: Metformin Tmax
Time Frame: Periods 1, 2, and 3 (before dosing, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 36 and 48 hours after dosing)
Population: All treated participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
hours | 4.78 (1.04) | 4.90 (1.13) | 4.11 (0.88)

18. Secondary Outcome: Metformin Fraction of AUC(0-inf) Contributed by AUC(0-t)(AUC[0-t]/AUC[0-inf])
Time Frame: Period 1 (before dosing, 0.167,0.25,0.5,0.75,1,1.5,2,3,4,5,6,7,8,10,12,18,24,36 and 48 hours after dosing)
Population: Treated participants (the smaller sample size for AUC(0-inf) was due to the inability to estimate Kel for some of the subjects).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 25 | 24 | 23
ratio | 0.979 (0.020) | 0.970 (0.026) | 0.965 (0.031)

19. Secondary Outcome: Safety: Adverse Events (AEs), Discontinuations Due to AEs, Deaths, and Serious AEs (SAEs)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: AEs: from initiation of study drug administration on Day 1/Period 1 through study discharge Day 3/Period 3. SAEs: from date of written consent until 30 days after discontinuation of dosing or participation in study if last scheduled visit occurred later.
Population: Safety Population = all participants who received any study drug.
Measure: Number; unit: Participants
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Number of Participants With At Least 1 AE | 3 | 2 | 4
  Discontinuation Due to an AE | 0 | 0 | 0
  Deaths | 0 | 0 | 0
  SAEs | 0 | 0 | 0

20. Secondary Outcome: Safety: Clinically Significant Laboratory, Vital Sign, Physical Examination, and Electrocardiogram (ECG) Abnormalities
Description: Abnormalities considered by the investigator to be clinically significant and/or reported as an AE.
Time Frame: From Day 1 of Period 1 through Day 3 of Period 3 (study discharge)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Treatment A - Saxagliptin + Metformin XR, Fed | Treatment B - FDC Tablet (Saxagliptin + Metformin XR), Fed | Treatment C - FDC Tablet (Saxagliptin + Metformin XR), Fasting
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Clinical Laboratory Abnormalities | 0 | 0 | 0
  Vital Sign Abnormalities | 0 | 0 | 0
  Physical Examination Abnormalities | 0 | 0 | 0
  12-Lead ECG Abnormalities | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Treatment A: 5 mg saxagliptin tablet + a single 500 mg metformin XR tablet under fed conditions
- Treatment C: FDC Tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fasting conditions
- Treatment B: Fixed-dose combination (FDC) tablet (5 mg Saxagliptin + 500 mg Metformin XR) under fed conditions
Arm/Group | Treatment A | Treatment C | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 4/30 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=30) | Treatment C (N=30) | Treatment B (N=30)
HEADACHE (Nervous system disorders) | 0 | 1 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1
LIP SWELLING (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.